CLINICAL TRIAL: NCT03524690
Title: Effects of Severe Negative Energy Balance on Inflammation During a Simulated Military Operation
Brief Title: Effects of Severe Negative Energy Balance on Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18-06HC
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized, cross-over controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUSOPS Balance (Active Comparator): Volunteers provided sufficient food to maintain energy balance.
  Interventions: Dietary Supplement: Energy Balance
- SUSOPS Negative Balance (Experimental): Volunteers provided insufficient food to maintain energy balance resulting in negative energy balance.
  Interventions: Dietary Supplement: Negative Energy Balance

INTERVENTIONS:
Dietary Supplement: Energy Balance — Energy Balance Sufficient food provided to maintain energy balance.
  Arms: SUSOPS Balance
Dietary Supplement: Negative Energy Balance — Negative Energy Balance Insufficient food provided to maintain energy balance resulting in negative energy balance.
  Arms: SUSOPS Negative Balance

SUMMARY:
The effects of prolonged negative energy balance, commonly observed in sustained military training and combat operations, on systemic inflammatory responses has not been determined. To define the putative role of energy balance on inflammation and its downstream effects, we will conduct a controlled laboratory study that simulates extensive physiological stressors to determine if inflammation is exacerbated by underfeeding. This design will test the hypothesis that maintaining energy balance will attenuate systemic inflammation and its potential negative effects on whole-body metabolic homeostasis in response to physiological stressors.

DETAILED DESCRIPTION:
Endurance exercise elicits skeletal muscle and systemic inflammation. Inflammation in response to endurance exercise is normally attenuated with adequate rest and recovery as skeletal muscle adapts with training. However, performing repeated bouts of prolonged and unaccustomed, muscle damaging (i.e., eccentric loading) endurance exercise may be detrimental to performance and limit the adaptive responses to exercise by diminishing the absorption of key nutrients. Warfighters are commonly exposed to such exercise bouts during sustained training and combat operations, the effects of which may be exacerbated by negative energy balance. Therefore, to define the putative role of energy balance on systemic inflammation, we will conduct a controlled laboratory study that simulates the physiological stressors imposed during sustained military training and combat operations to determine if systemic inflammation is exacerbated by underfeeding.

Twenty-six male, non-obese (body mass index 19.9-29.9 kg/m2), physically active adults will be recruited to participate in a 32 d, longitudinal study. The study is comprised of four sequential phases: 1) a 96 h testing period, 2) a 7 day recovery period (Recovery 1), 3) a second, 96 h testing period, and 4) a 14 d recovery period (Recovery 2). During testing, subjects will be randomized to consume either sufficient food (combat rations) to maintain energy balance or will be provided a restricted amount of food to elicit severe negative energy balance. Mineral absorption studies and will be conducted during each testing condition, energy balance and energy negative balance. This design will test the hypothesis that maintaining energy balance will attenuate systemic inflammation and its potential negative effects on whole-body metabolic homeostasis in response to physiological stressors.

ELIGIBILITY:
Inclusion Criteria:

* Men who are active duty military, aged 18 - 39 years
* Weight stable in the past 2 months (± 2.27 kg)
* Healthy without evidence of chronic illness, medication use, or musculoskeletal injury as determined by the USARIEM Office of Medical Support and Oversight (OMSO)
* Recreationally active (2-4 days per week aerobic and/or resistance exercise)
* Refrain from taking any pain-relievers (e.g., acetaminophen), nonsteroidal anti-inflammatory drugs (e.g., aspirin, Advil®, Aleve®, Naprosyn®), or any other aspirin-containing product for 10 days before starting and at least 5 days after completing the study
* Refrain from the use of alcohol and nicotine for the duration of the study
* Willing to refrain from alcohol, smoking any nicotine product (includes e-cigarettes), vaping, chewing tobacco, caffeine, and dietary supplement use, and from consumption of probiotic-containing foods (e.g., yogurt) throughout the entire study period (vitamin/mineral supplements cannot be taken for at least 2 weeks before starting the study)
* Supervisor approval for non-HRV Active Duty Military working within the US Army Natick Soldier Systems Center
* Reports having a bowel movement at least as frequently as every-other-day

Exclusion Criteria:

* Musculoskeletal injuries that compromise exercise capability
* Metabolic or cardiovascular abnormalities (e.g., kidney disease, diabetes, cardiovascular disease, etc.)
* History of any disease or abnormality of the gastrointestinal tract including (but not limited to) diverticulosis, diverticulitis and inflammatory bowel disease, peptic ulcer disease, Crohn's disease, ulcerative colitis; or previous gastrointestinal surgery
* Anemic (plasma ferritin < 40 µg/L, hemoglobin < 13 g/dL) and Sickle Cell Anemia/Trait
* C-reactive protein (CRP) > 5 mg/dL
* Abnormal PT/PTT test or problems with blood clotting
* History of complications with lidocaine
* Evidence of any physical, mental, and/or medical conditions that would make the proposed studies relatively more hazardous as determined by OMSO
* Present condition of alcoholism or other substance abuse issues; use of anabolic steroids
* Blood donation within 4 months of beginning the study
* Oral antibiotic use within 3 months of participation
* Colonoscopy within 3 months of participation
* Use of laxatives, stool softeners, or anti-diarrheal medications more than once/month
* Currently using benzodiazepines, anti-depressants or anti-histamines
* Pacemaker or other implanted electronic medical device
* Are unwilling or unable to eat study diets and foods provided and/or follow exercise prescriptions

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
The effects of a simulated military operation on systemic inflammation | 6 hour measure
  Assessed using blood assays.

SECONDARY OUTCOMES:
The effects of energy balance and severe energy deficit on inflammation during a simulated military operation | 6 hour measure
  Assessed using mineral absorption from stable isotopes.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan M Pasiakos, PhD, Principal Investigator — Military Nutrition Division, USARIEM
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hennigar SR, McClung JP, Hatch-McChesney A, Allen JT, Wilson MA, Carrigan CT, Murphy NE, Teien HK, Martini S, Gwin JA, Karl JP, Margolis LM, Pasiakos SM. Energy deficit increases hepcidin and exacerbates declines in dietary iron absorption following strenuous physical activity: a randomized-controlled cross-over trial. Am J Clin Nutr. 2021 Feb 2;113(2):359-369. doi: 10.1093/ajcn/nqaa289. PMID 33184627

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03524690/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT03524690/ICF_001.pdf